CLINICAL TRIAL: NCT01534975
Title: A Prospective, Single-Center Double-Blind Randomized Study in Subjects Undergoing Coronary Computed Tomography Angiography (CCTA) Examination (VISIPAQUE Randomized Study)
Brief Title: Comparison of Contrast Agents During CT Angiography
Acronym: Visipaque
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center (Other)
Collaborators: General Electric (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: Visipaque
Record Dates: First submitted 2012-02-14; First posted 2012-02-17 (Estimated); Results first posted 2018-03-01 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2017-03

CONDITIONS: Contrast Enhancement on Cardiac CT
Keywords: cardiac CT; enhancement; contrast; safety; image quality

STUDY DESIGN:
Intervention Model Description: randomized cohort into 4 groups - each group with a different contrast agent (omnipaque, visipaque 280, visipaque 320, isovue)
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Iodixanol 320 (Active Comparator): group 1 will receive iodixanol 320 as the contrast agent during CT acquisition. this will reflect the "intervention" of that arm, by testing the diagnostic ability of this contrast agent to perform cardiac CT angiography
  Interventions: Diagnostic Test: contrast agent
- iohexol 350 (Active Comparator): group 2 will receive iohexol 350 as the contrast agent during CT acquisition. this will reflect the "intervention" of that arm, by testing the diagnostic ability of this contrast agent to perform cardiac CT angiography
  Interventions: Diagnostic Test: contrast agent
- iopamidol 370 (Active Comparator): group 3 will receive iopamidol 370 as the contrast agent during CT acquisition. this will reflect the "intervention" of that arm, by testing the diagnostic ability of this contrast agent to perform cardiac CT angiography
  Interventions: Diagnostic Test: contrast agent
- iodixanol 270 (Active Comparator): group 4 will receive iodixanol 270 as the contrast agent during CT acquisition. this will reflect the "intervention" of that arm, by testing the diagnostic ability of this contrast agent to perform cardiac CT angiography
  Interventions: Diagnostic Test: contrast agent

INTERVENTIONS:
Diagnostic Test: contrast agent — we are randomizing patients to different contrast agents.

SUMMARY:
The purpose of this study is to compare the effects of a certain contrast agent (iodixanol) to two other commonly used contrast agents called Iopamidol (Isovue) and iohexol (Omnipaque), on heart and kidney safety in patients undergoing a cardiac CT angiogram. The investigators will evaluate whether iodixanol 320 (Visipaque®), an iso-osmolar agent, is better tolerated (flushing, injection site pain/warmth, headache, nausea) and provides equal image quality compared with iohexol 350 (Omnipaque®) and Isovue 370 during 64-slice multidetector computed tomography angiography (MDCTA). A fourth group (Visipaque 270) will be included, using low radiation dose technology during acquisition, to evaluate image quality, tolerability, and contrast enhancement compared to both Visipaque 320 and Omnipaque and Isovue. In addition to image quality, tolerability, and contrast enhancement, the investigators will evaluate heart rate, adverse events, reimaging, costs, and patient satisfaction among all four cohorts.

The study will recruit 400 participants already undergoing CT angiography and consent and randomize them to one of four groups. Each of the possible contrast agents used are commonly used for CT angiography, so the primary risk is loss of confidentiality and being asked questions about tolerability. All other facets of the study (3 lead ECG, beta blockade, nitroglycerine use, CT angiography and contrast administration) are standard of care and being done for clinical uses.

DETAILED DESCRIPTION:
CTA infusion is administered using a 5 ml/sec IV iodinated contrast infusion. 50-70 ml of iodinated contrast is used for the scan depending on the patient's body habitus. The total contrast dose must not exceed 70 ml. An automated bolus tracking feature (SmartPrep, GE Healthcare, Milwaukee, USA) is used to judge contrast bolus arrival and optimize image quality. Patients will be asked to hold their breaths during scanning for up to 10 seconds. A Field of View (FOV) of 25 cm is adjusted to include the heart from below the carina to just below diaphragm. The aorta will be included in the FOV to exclude aortic pathology (ie. dissection, aneurysm, etc.). For patients in sinus rhythm, prospective ECG gating centered at 75% of the R-R interval is used while those in Atrial fibrillation or HR >65 despite oral and IV medications, a retrospective gating is used. The following parameters are used Tube voltage = 100-120kV (based on body habitus), tube current = 400 mA, gantry rotation speed = 0.35 seconds, slice thickness = 0.625 mm, rows = 64, coverage = 128-160 mm.

Estimated radiation dose is = 2-5 mSv dependent on BMI, cardiac height and heart rate. A post acquisition software (Adaptive Statistical Iterative Reconstruction, GE healthcare, Milwaukee, USA) is used to reduce pixel noise standard deviation (noise) by 30 percent and allows for reduced mA in the acquisition while still yielding diagnostic images, thereby reducing total dose required. At the conclusion of each acquisition, technologists collect a survey of patient satisfaction quantifying side effects of different contrasts: flushing, headache, nausea, and pain at injection site as mild, moderate or severe.

Advantage Workstation 4.6 software (GE healthcare, Milwaukee, USA) is used for post acquisition processing. Readers, who are blinded to the type of contrast media used, assess image quality by measuring contrast enhancement in aorta, LV myocardium, left main, proximal Left Anterior Descending artery, proximal and distal Right Coronary arteries. Subjects with coronary artery bypass graft and stents are excluded. Heart rate (HR) variability during the scan is also evaluated. A comparison of the degree of contrast enhancement of the coronary lumen as well as the differences for each of the four contrast agents will be measured and reported, stratified by 100 kVp and 120 kVp acquisition. The image quality of 17 coronary artery segments will be graded by two cardiologists in consensus with the use of a four-point scale (1= excellent, 2=good, 3=fair , 4= poor enhancement) blinded to contrast agent administration.

Statistical Analysis:

All analysis is conducted using SPSS 18.0 for window (SPSS Inc., Chicago, IL, USA). Comparisons between groups are performed using a Student t-test for continuous variables with normal distributions and the Mann-Whitney U test for continuous variables with non-normal distributions. Categorical variables were analyzed by means of χ2 analysis. Correlation between minimum HR and maximum HR was calculated with the Pearson correlation coefficient. The Cochran-Mantel-Haenszel test was used for analyzing the difference in visual quality between two groups.

ELIGIBILITY:
Inclusion Criteria:

Subjects may be included in the study if they meet all of the following criteria:

1. The subject is over 18 years old.
2. Subject scheduled to undergo a contrast-enhanced CCTA examination
3. The subject has no contra-indication to receiving iodinated contrast administration (allergy, renal insufficiency).
4. The subject has provided signed and dated informed consent

Exclusion criteria:

Subjects must be excluded from participating in this study if they meet the following criteria:

1. Subjects have known contra-indication to contrast administration:

   * Renal insufficiency as defined by GFR < 50
   * Known contrast allergy
2. Pregnant or possibly pregnant subjects will be excluded -Women of childbearing potential will undergo urine pregnancy test prior to CT scanning.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 513 (Actual)
Dates: Start 2012-01; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Los Angeles Biomedical Research Institute, Torrance, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Honoris L, Zhong Y, Chu E, Rosenthal D, Li D, Lam F, Budoff MJ. Comparison of contrast enhancement, image quality and tolerability in Coronary CT angiography using 4 contrast agents: A prospective randomized trial. Int J Cardiol. 2015;186:126-8. doi: 10.1016/j.ijcard.2015.03.240. Epub 2015 Mar 19. No abstract available. PMID 25818754

RESULTS

PARTICIPANT FLOW:
Groups:
- Iodixanol 320: group 1 Iodixanol 320
- Iohexol 350: group 2 iohexol 350
- Iopamidol 370: group 3 iopamidol 370
- Iodixanol 270: group 4 iodixanol 270
Period: Overall Study
Arm/Group | Iodixanol 320 | Iohexol 350 | Iopamidol 370 | Iodixanol 270
Started | 136 | 133 | 160 | 84
Completed | 136 | 133 | 160 | 84
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Iodixanol 320 | Iohexol 350 | Iopamidol 370 | Iodixanol 270 | Total
Number analyzed (Participants) | 136 | 133 | 160 | 84 | 513
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 92 | 90 | 110 | 60 | 352
  >=65 years | 44 | 43 | 50 | 24 | 161
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (11.7) | 62.3 (11.4) | 61.4 (10.8) | 60.4 (11.2) | 62 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66 | 63 | 76 | 40 | 245
  Male | 70 | 70 | 84 | 44 | 268
Region of Enrollment [Number; unit: participants]
  United States | 136 | 133 | 160 | 84 | 513

OUTCOME MEASURES:

1. Primary Outcome: Image Quality of the CT Scans Using Different Contrast Agents
Description: Attenuation (HU) in the ascending aorta, standard deviation (SD) of aorta, will be measured,.
Time Frame: 1 year
Measure: Mean (Standard Deviation); unit: hounsfield units
Groups:
- Iodixanol 320: group 1
- Iohexol 350: group 2
- Iopamidol 370: group 3
- Iodixanol 270: group 4
Arm/Group | Iodixanol 320 | Iohexol 350 | Iopamidol 370 | Iodixanol 270
Number analyzed (Participants) | 136 | 133 | 160 | 84
hounsfield units | 333 (59) | 357 (64) | 362 (68) | 288 (61)

ADVERSE EVENTS:
Arm/Group | Iodixanol 320 | Iohexol 350 | Iopamidol 370 | Iodixanol 270
Serious Adverse Events (participants affected / at risk) | 0/136 | 0/133 | 0/160 | 0/84
Other Adverse Events (participants affected / at risk) | 98/136 | 122/133 | 152/160 | 52/84
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Iodixanol 320 (N=136) | Iohexol 350 (N=133) | Iopamidol 370 (N=160) | Iodixanol 270 (N=84)
flushing (Blood and lymphatic system disorders) | 98 (98) | 122 (122) | 152 (152) | 52 (52) — patients reported flushing after administration of contrast

LIMITATIONS AND CAVEATS:
study was performed as outlined, sample sizes are appropriate, there were no technical problems.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No